CLINICAL TRIAL: NCT03756506
Title: An Evaluation of the Use of a Novel Microbicidal Liquid Polymer for the Reduction of Pin-tract Infection in Research Participants Receiving External Fixation Following Deformity Correction and Traumatic Provisional Fixation
Brief Title: The Use of a Novel Microbicidal Liquid Polymer for the Reduction of Pin Track Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prevent-Plus LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-01
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Results first posted 2020-07-13 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2020-06

CONDITIONS: Infection; Post-operative Care
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: The study will enroll 12 total research participants (6 control research participants and 6 research participants) with approximately 120 pin sites (approximately 60 in the Control group and 60 in the DuraDerm® group). Each research participant undergoing Deformity Correction and/or Traumatic Provisional Surgery will be asked to participate in the study to evaluate if the topical application of a Novel Microbicidal Liquid Polymer as an additional step in the management of post-operative pin track site care reduces the incidence of pin track infections. Investigational Review Board (IRB) approval will be obtained and informed research participant consent will be obtained from each research participant.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Novel Microbicidal Liquid Polymer (Active Comparator): All pins and wire sites will be cleaned daily while hospitalized. Basic pin care will be performed once daily by hospital nursing staff prior to discharge. Following discharge from the hospital, the pin care protocol will be continued by research participant's caregiver.Research participants will be instructed to notify the Principal Investigator if they observe any signs or symptoms of infection. These include redness around pin site, discharge,tenderness in the soft tissue, loosening of the pin, nausea, vomiting, fever or chills.
  Step 1: Brush the pin sites with saline using an ordinary soft toothbrush or gauze with sterile gloves Step 2: If following Step 1, debris remains, use forceps (tweezers) to gently remove debris. Step 3: Apply product with Q-tip on clean dry wound around (extending approximately one inch around pin site) and on the pin. The Polymer will be applied daily while in the hospital and then at a minimum of at least three times a week until pin removal.
  Interventions: Device: Novel Microbicidal Liquid Polymer
- Control group: no Novel Microbicidal Liquid Polymer (No Intervention): The usual care of pin track sites will be followed as outlined belowAll pins and wire sites will be cleaned daily while hospitalized. Basic pin care will be performed once daily by hospital nursing staff prior to discharge. Following discharge from the hospital, the pin care protocol will be continued by research participant's caregiver.
  Research participants will be instructed to notify the Principal Investigator if they observe any signs or symptoms of infection. These include redness around pin site, discharge, tenderness in the soft tissue, loosening of the pin, nausea, vomiting, fever or chills.
  Research participants will be instructed that the approach to pin care should occur in a step-wise fashion. Step 1: Brush the pin sites with saline using an ordinary soft toothbrush or gauze with sterile gloves Step 2: If following Step 1, debris remains, use forceps (tweezers) to gently remove debris.

INTERVENTIONS:
Device: Novel Microbicidal Liquid Polymer — The polymer is a 510K FDA cleared medical device indicated for providing a covering over minor wounds and scrapes that are clean and dry. The microbicidal liquid solution consists of organic polymers . The unique formulation eradicates any organisms (bacteria, fungi, viruses) it comes in contact with. This is a result of the solvent's activity against an infinite number of organisms After eradication is complete, the solvent then transitions into a clear, elastomeric, non-odorous film for covering disrupted tissue. The film protects the wound against entry of water, dirt, and germs. The film is elastomeric and protects in difficult regions where flexing, bending and creasing skin occurs. The clear film forms in less than a minute.6 DuraDerm® should not be used to the treat deep infected wounds. DuraDerm® can be used to protect disrupted skin surface of wounds that are clean and dry.
  Arms: Novel Microbicidal Liquid Polymer

SUMMARY:
The purpose of the study is to investigate additional clinical uses for the polymer, which is a FDA approved, 510k, medical device, but has not been approved for use on patients with pin track sites as a way to lower the infection rate and is investigational for this purpose. The approved uses include wound care and post-operative care.

About 13 subjects will take part in this study.

DETAILED DESCRIPTION:
Study Objectives Research participants eligible for the study will be those undergoing Deformity Correction and Traumatic Provisional Fixation. These research participants have a number of pins placed to ensure this required rigid fixation. The number of external fixation pins averages approximately ten per research participant.

It is a 510K FDA cleared medical device indicated for providing a covering over minor wounds and scrapes that are clean and dry. The microbicidal liquid solution consists of organic polymer dissolved in methylene chloride organic solvent. The unique formulation eradicates any organisms (bacteria, fungi, viruses) it comes in contact with. This is a result of the methylene chloride's activity against an infinite number of organisms. The methylene chloride evaporates leaving a clear, elastomeric, non-odorous film for covering minor wounds. The film protects the wound against entry of water, dirt, and germs. The film is elastomeric and protects in difficult regions where flexing, bending and creasing skin occurs. The clear film forms in less than a minute. Application is commonly accomplished using a cotton tip applicator. The liquid is applied on and around the wound extending at least an inch and a quarter beyond the edges of the wound. Momentary stinging may occur upon initial application. The film commonly remains intact for one to three days or longer depending on exposure to rubbing, flexing, or soap and water. This film is resistant to degradation by water alone, but can be easily removed with the combination of soap and water or it can be gently peeled off starting at the outer edges. It is for external use only. It is not intended for use on deep or infected wounds or puncture wounds, or for use near the eyes, mouth, or nose. Intentional inhaling of the contents may be harmful or fatal. The bottle should be tightly capped after each use to prevent evaporation of the solvent.7

This Principle Investigator has previously utilized and topically applied the product as an additional step in the treatment protocol for pin site care for several reconstructive surgery patients (approximately 25) with over 200 pin sites with only 2 pin site infections. This represents a significant reduction from the average incidence of pin site infections reported in the literature (<1% vs 27% on a per research participant basis). A recently published retrospective case series evaluating this microbicidal polymer dressing reported 6 patients and 66 pins had no infections when Duraderm® was used as part of their pin site care regimen.8

This study was undertaken to formally evaluate whether this microbial liquid po used on pin sites leads to a reduction in pin track infections when compared to a control group as well as the reported average incidence in the literature.

ELIGIBILITY:
Inclusion Criteria:

1. Deformity correction, traumatic provisional fixation
2. All pin sites are stable
3. 18 years of age or greater
4. No known contraindication to receive product

Exclusion Criteria:

1. Age less than 18 years
2. Known allergy to Methylene Chloride
3. Known sensitivity to organic polymers
4. Non-clean, dry wound at pin
5. Vulnerable research participants (Institutionalized, students, employees, prisoners, or those with decisional incapacity, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shital Pema, DPM, Principal Investigator — Kettering Health System
Locations (1):
- Julie Morris, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: dlk
Groups:
- DuraDerm® Group: All pins and wire sites will be cleaned daily while hospitalized. Basic pin care will be performed once daily by hospital nursing staff prior to discharge. Following discharge from the hospital, the pin care protocol will be continued by research participant's caregiver.Research participants will be instructed to notify the Principal Investigator if they observe any signs or symptoms of infection. These include redness around pin site, discharge,tenderness in the soft tissue, loosening of the pin, nausea, vomiting, fever or chills.
  Step 1: Brush the pin sites with saline using an ordinary soft toothbrush or gauze with sterile gloves Step 2: If following Step 1, debris remains, use forceps (tweezers) to gently remove debris. Step 3: Apply DuraDerm® with Q-tip on clean dry wound around (extending approximately one inch around pin site) and on the pin. DuraDerm® will be applied daily while in the hospital and then at a minimum of at least three times a week until pin removal.
- Control Group: no DuraDerm: The usual care of pin track sites will be followed as outlined belowAll pins and wire sites will be cleaned daily while hospitalized. Basic pin care will be performed once daily by hospital nursing staff prior to discharge. Following discharge from the hospital, the pin care protocol will be continued by research participant's caregiver.
  Research participants will be instructed to notify the Principal Investigator if they observe any signs or symptoms of infection. These include redness around pin site, discharge, tenderness in the soft tissue, loosening of the pin, nausea, vomiting, fever or chills.
  Research participants will be instructed that the approach to pin care should occur in a step-wise fashion. Step 1: Brush the pin sites with saline using an ordinary soft toothbrush or gauze with sterile gloves Step 2: If following Step 1, debris remains, use forceps (tweezers) to gently remove debris.
Period: Overall Study
Arm/Group | DuraDerm® Group | Control Group: no DuraDerm
Started | 7 | 6
Completed | 6 | 6
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- DuraDerm® Group: All pins and wire sites will be cleaned daily while hospitalized. Basic pin care will be performed once daily by hospital nursing staff prior to discharge.
  Step 1: Brush the pin sites with saline using an ordinary soft toothbrush or gauze with sterile gloves Step 2: If following Step 1, debris remains, use forceps (tweezers) to gently remove debris. Step 3: Apply DuraDerm® with Q-tip on clean dry wound around (extending approximately one inch around pin site) and on the pin. DuraDerm® will be applied daily while in the hospital and then at a minimum of at least three times a week until pin removal.
- Control Group: no DuraDerm: The usual care of pin track sites will be followed as outlined below. All pins and wire sites will be cleaned daily while hospitalized. Basic pin care will be performed once daily by hospital nursing staff prior to discharge. Following discharge from the hospital, the pin care protocol will be continued by research participant's caregiver.
  Research participants will be instructed to notify the Principal Investigator if they observe any signs or symptoms of infection. These include redness around pin site, discharge, tenderness in the soft tissue, loosening of the pin, nausea, vomiting, fever or chills.
  Research participants will be instructed that the approach to pin care should occur in a step-wise fashion. Step 1: Brush the pin sites with saline using an ordinary soft toothbrush or gauze with sterile gloves Step 2: If following Step 1, debris remains, use forceps (tweezers) to gently remove debris.
- Total: Total of all reporting groups
Arm/Group | DuraDerm® Group | Control Group: no DuraDerm | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pin Track Infection Rate Among Research Participants Based on Number of Pins Undergoing Deformity Correction and Traumatic Provisional Fixation
Description: Research participants identified for the study will be those undergoing Deformity Correction and Traumatic Provisional Fixation who are under the care of the Primary Investigator. These research participants have a number of pins placed to ensure this required rigid fixation. The number of external fixation pins averages approximately ten per research participant. Research participants seen by the Primary Investigator who will be undergoing deformity correction or traumatic provisional fixation, will be invited to take part in this research study. No recruitment of the Principal Investigator's own students, employees, or family members will be allowed. Research participants who do not wish to participate in this randomized study will be provided the standard pin track care protocol this investigator utilizes for his research participants and will not have the opportunity to receive DuraDerm®.
Time Frame: 10 months
Population: Infection rate was analyzed on a per patient and a per pin basis.
Measure: Count of Units; unit: Pins
Units Other Than Participants: Pins
Groups:
- DuraDerm® Patient Group: All pins and wire sites will be cleaned daily while hospitalized. Basic pin care will be performed once daily by hospital nursing staff prior to discharge. Following discharge from the hospital, the pin care protocol will be continued by research participant's caregiver.Research participants will be instructed to notify the Principal Investigator if they observe any signs or symptoms of infection. These include redness around pin site, discharge,tenderness in the soft tissue, loosening of the pin, nausea, vomiting, fever or chills.
  Step 1: Brush the pin sites with saline using an ordinary soft toothbrush or gauze with sterile gloves Step 2: If following Step 1, debris remains, use forceps (tweezers) to gently remove debris. Step 3: Apply DuraDerm® with Q-tip on clean dry wound around (extending approximately one inch around pin site) and on the pin. DuraDerm® will be applied daily while in the hospital and then at a minimum of at least three times a week until pin removal.
- Patient Control Group: no DuraDerm: The usual care of pin track sites will be followed as outlined belowAll pins and wire sites will be cleaned daily while hospitalized. Basic pin care will be performed once daily by hospital nursing staff prior to discharge. Following discharge from the hospital, the pin care protocol will be continued by research participant's caregiver.
  Research participants will be instructed to notify the Principal Investigator if they observe any signs or symptoms of infection. These include redness around pin site, discharge, tenderness in the soft tissue, loosening of the pin, nausea, vomiting, fever or chills.
  Research participants will be instructed that the approach to pin care should occur in a step-wise fashion. Step 1: Brush the pin sites with saline using an ordinary soft toothbrush or gauze with sterile gloves Step 2: If following Step 1, debris remains, use forceps (tweezers) to gently remove debris.
Arm/Group | DuraDerm® Patient Group | Patient Control Group: no DuraDerm
Number analyzed (Participants) | 6 | 6
Number analyzed (Pins) | 60 | 60
Pins | 0 | 14

2. Primary Outcome: Pin Track Infection Rate Among Research Participants Undergoing Deformity Correction and Traumatic Provisional Fixation
Description: as for outcome 1
Time Frame: 10 months
Population: Infection rate was analyzed on a per patient basis.
Measure: Count of Participants; unit: Participants
Arm/Group | DuraDerm® Patient Group | Patient Control Group: no DuraDerm
Number analyzed (Participants) | 6 | 6
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 4-8 weeks depending on patient's length of pin placement.
Arm/Group | DuraDerm® Group | Control Group: no DuraDerm
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
This study is limited by its sample size when evaluating infection rate on a per patient basis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT03756506/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT03756506/SAP_002.pdf